CLINICAL TRIAL: NCT03397498
Title: Computerized Cognitive Intervention in the Oldest-Old: A Feasibility Study
Brief Title: Computerized Cognitive Intervention in the Oldest-Old
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 09-2339
Record Dates: First submitted 2018-01-05; First posted 2018-01-12 (Actual); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Cognition; Dementia
Keywords: computerized cognitive training
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants are not told which group they are assigned to, and the investigator (PI) and coordinators completing the cognitive evaluation are not told which group the participants are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Computerized cognitive training (Experimental): Received the Computerized cognitive training program, CogniFit™
  Interventions: Behavioral: CogniFit™
- Control-games (Active Comparator): Received the Computerized games program
  Interventions: Behavioral: Control-games

INTERVENTIONS:
Behavioral: CogniFit™ — The program utilizes 21 tasks, which may develop 14 cognitive domains: awareness, inhibition, spatial perception, visual short term memory, working memory, hand-eye coordination, visual scanning, response time, divided attention, time estimation, visual perception, shifting, naming, and planning.
  Other Names: Computerized cognitive training program
  Arms: Computerized cognitive training
Behavioral: Control-games — The program utilizes classic computer games, which may develop cognitive domains. Games will be used over 8 weeks. The participants will use the program 3 days a week, with one rest day between each session. Each session lasts approximately 20 minutes. The participant will use the program for a total number of 24 sessions.
  Other Names: Computerized games program
  Arms: Control-games

SUMMARY:
Little is known about preventive strategies with immediate public health impact for cognitive functioning in the oldest-old (OO). Cognitive training improves cognitive functioning in the young-old (YO; 60 to 84), yet has not been examined in the OO.

Clinical trials are needed to determine if computerized cognitive training is effective at preventing or delaying cognitive decline in the OO. In order to develop such trials, information regarding use of computers and internet by the OO, and the ability and interest in such a program, must be determined.

This study will examine the effects of a computerized cognitive training program, CogniFit™, with a "classic" computerized games program, on cognitive functioning in cognitively healthy OO subjects. Information regarding use of computers and internet by the OO will be collected. Interest in and ability to complete a computerized cognitive training program will be examined, along with the cognitive, demographic, biological, and lifestyle characteristics related to this interest and ability.

Efficacy of the CogniFit™ and games programs will be assessed immediately following the training and four months after completing the training. The researchers expect that those who use the CogniFit™ program will have greater improvements than those using the games program. Finally, the participants' characteristics related to the efficacy of the programs will be examined.

Subjects recruited for this project will include those already participating in several studies of aging and cognition at the Mount Sinai School of Medicine. Recruiting from this pool of subjects will provide this program with baseline information regarding numerous subject characteristics, including cognition, family history, lifestyle, and cardiovascular information.

This study will inform future large-scale clinical trials of computerized cognitive training programs in the elderly, as well as provide information regarding the efficacy of such training in the OO. In addition, the study will identify characteristics affecting efficacy of computerized training, and thus, may suggest mechanisms through which cognitive training improves cognitive functioning in the most senior citizens of our society.

DETAILED DESCRIPTION:
Specific Aim 1- To estimate, in cognitively normal OO, rates of 1) computer and internet use, 2) willingness to participate in a computerized cognitive training program, 3) ability to comply with the program to its completion.

Specific Aim 1a- To explore the relationships of baseline global cognition, sociodemographic, ADL/IADL, lifestyle, and biological characteristics with willingness to participate in, and with completion of a computerized cognitive training program.

Specific aim 2 - To compare the effectiveness of the CogniFit. and games programs 2 months after initiation of the intervention (corresponding to the time to complete the intervention).

Specific aim 2a - To compare the effectiveness of the CogniFit. and games programs 6 months after initiation of intervention Specific aim 3- To explore the relevance of the wide range of already available sociodemographic, lifestyle, ADL/IADL, and biological characteristics of subjects with the differential effectiveness of the programs.

Results of this study will provide essential information for planning a large-scale trial of computerized cognitive training program for the OO.

The current lack of disease modifying treatment to delay onset of slow progression to Alzheimer's disease (AD), and the robust epidemiologic evidence suggesting modifiable protective life-style factors (eg. cognitive and physical activity have led to particular interest in life-style interventions that delay the onset or slow the progression of cognitive decline.

ELIGIBILITY:
Inclusion Criteria:

* Age 80+
* Normal cognition by consensus conference, MMSE> 25th percentile norm, CDR=0
* Has computer with internet access that is capable of running the computerized cognitive training program.
* Willing to dedicate the necessary time to the project

Exclusion Criteria:

* Prior or current participation in another cognitive intervention study
* Medical disease that precludes consistent participation or that affects cognition
* Poor vision
* Poor hearing

Min Age: 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-03-10 (Actual); Primary Completion 2014-12-16 (Actual); Study Completion 2014-12-16 (Actual)

PRIMARY OUTCOMES:
Change in Global Cognition Composite | Baseline and after completion of program (approximately 7-8 weeks)
  Memory, Immediate recall; Word List Memory, Delayed recall; Word List Memory, Recognition; Logical Memory Story A, Immediate recall; Logical Memory Story A, Delayed recall; Logical Memory Story A, Recognition, Target Cancellation Tests (diamond and TMX); Trail Making Test (Parts A and B); Digit Symbol Substitution Test; Digit Span tests (Forward and Backward), Similarities; Boston Naming Test; and Category Fluency and Letter Fluency tests at completion of program as compared to baseline.

SECONDARY OUTCOMES:
Change in Memory Function | Baseline and after completion of program (approximately 7-8 weeks)
  A 10-item word list is presented over 3 trials (at the rate of 1 every 2 seconds) with a different word order each trial. The participant reads each word aloud as it is presented and then asked to recall as many words as possible. The range is 0 - 10 for each trial, with a Trial Total of 30. After a short delay the participant is asked to recall as many of the 10 words as they can. Word List Recognition: Immediately after the Delayed Recall task, the participant is asked to identify the 10 words from the list of target words and ten distractor words. There is a max of 10 correct 'Yes' responses and 10 correct 'No' responses. To adjust for chance, the score is calculated as the total number of correct answers minus 10. A Savings score is calculated to reflect the ability to recall learned information after a delay; this score is obtained by dividing the number of words recalled after the delay by the total number correct on Trial 3 and compared at completion of program to baseline.
Change in Logical Memory Story A | Baseline and after completion of program (approximately 7-8 weeks)
  The LM subtest of the WMS-R is a standardized assessment of narrative episodic memory. A short story is orally presented, and the examinee is asked to recall the story verbatim (immediate recall). Approximately 20 or 30 min later, free recall of the story is again elicited (delayed recall). at completion of program as compared to baseline.
Change in Attention/Executive function score | Baseline and after completion of program (approximately 7-8 weeks)
  Attention/Executive function score - composite of Target Cancellation Tests (diamond and TMX); Trail Making Test (Parts A and B); Digit Symbol Substitution Test; and Digit Span tests (Forward and Backward) at completion of program as compared to baseline.
Change in Language function score | Baseline and after completion of program (approximately 7-8 weeks)
  Language function score - composite of Similarities; Boston Naming Test; and Category Fluency and Letter Fluency tests at completion of program as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Michal Schnaider-Beeri, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Jewish Home Lifecare, New York, New York
  - Icahn School of Medicine at Mount Sinia, New York, New York